CLINICAL TRIAL: NCT06463405
Title: Patient Perception and Oral Function of Implant-supported Restorations Replacing Posterior Teeth
Brief Title: Patient Perception and Oral Function of Implant Restorations
Acronym: REPLACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Klaus Gotfredsen, Professor, University of Copenhagen
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: REPLACE
Record Dates: First submitted 2024-05-30; First posted 2024-06-17 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Dental Occlusion
Keywords: Removable Partial Dentures; Dental Implants; Jaw relation record
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Splinted implant restorations (Other)
  Interventions: Other: Splinted
- Non-splinted implant restorations (Other)
  Interventions: Other: Splinted

INTERVENTIONS:
Other: Splinted — The investigators will compare splinted versus non-splinted crowns in a randomized design. Whether the crowns will be splinted or not are decided by distant randomization separate from clinicians conducting the trial. Twenty sealed envelopes will be opened where its stands whether the crowns has to be splinted crowns or non-splinted crowns. The implants in the splinted side will have an intermediate titanium abutment and impression will be taken at abutment level, whereas impressions in the non-splinted side will be taken directly at the fixture level. The splinted as well as the non-splinted crowns will be screw-retained and produced in monolithic zirconia. An open-tray technique / (scanning) will be used for both reconstructions.
  Other Names: Non-splinted

SUMMARY:
The overall aim is to evaluate the patient-reported outcome and efficiency of replacing posterior teeth with implant-supported crowns compared to RDPs and no treatment. Sub-aims are to evaluate a new 3D-methods for registration of occlusion and to test two crown designs.

Thus, the study design has three aims:

* To analyze patient perception including OHRQoL, when missing posterior teeth are replaced with implant-supported crowns compared to removable dental prostheses (RDPs) or no replacement.
* To develop and validate new 3D digital methods for assessing occlusal contacts between upper and lower jaw and to analyze the methods relation to masticatory ability and efficiency.
* To compare the difference in biological technical outcomes between splinted and non-splinted implant-supported crowns over time.

DETAILED DESCRIPTION:
Hypotheses

* No difference in patient perception of mastication and OHRQoL between no treatment, RDPs and implant-supported crowns in the posterior region
* No difference between two different digital techniques (T-scan and 3D Intraoral scanning) in measuring the occlusal contact points and area.
* No difference in biological and technical outcomes between splinted and non-splinted implant-supported crowns

Material and methods. Participants Partially edentulous subjects with missing posterior teeth (Kennedy class I or class II) in the upper or lower jaw, in need for fixed implant-supported crowns to replace the missing teeth are offered to be enrolled if they fulfill the following inclusion criteria. The participants must be in good health and with no contraindications for undergoing dento-alveolar surgery.

Subjects presenting with the following conditions will be excluded from the study:

* Untreated or active, progressive periodontitis
* Intake of (high dose) antiresorptive medicine or earlier medication related osteonecrosis of the jaw
* Therapeutic radiation to the head and neck
* Uncontrolled diabetes or systemic corticosteroids
* Heavy smoking (>20 cigarettes/day)
* An inability to open the mouth wide enough to place implants
* Decayed or unrestored anterior/premolar teeth
* Need for major bone augmentation (e.g., bone block graft, extensive augmentations with second operation for implant insertion)
* < 8 mm bone height to the alveolar nerve or sinus maxillaris
* Parafunctional habits or untreated temporomandibular dysfunctions or orofacial pain
* Unable to cooperate or too ill to complete the experiment
* Lack of signed informed consent A participant, who no longer wishes to participate in the trial, can withdraw her/his informed consent at any time. Withdrawn subjects can give information of which aspects of the trial she/he wishes to withdraw from.

All included subjects must have a natural dentition or fixed implant-supported reconstructions in the opposite jaw of at least two premolar equivalents occluding against the planned implant-supported crowns. If the teeth in the opposing jaw are elongated a coronal reduction will be performed to create unequivocally occlusal plane.

Free-end dentitions with missing teeth behind the canine, 1 or 2 premolars can be included. Patients from the dental school as well as patients from private practice will be invited to participate in the study when funding is achieved.

Pre-examinations and methods Participants will be pre-examined to be sure the inclusion and exclusion criteria is full filled (Figure 1). A Panoramic X-ray will be used to screen the tooth- and periodontal status. If these are full-filled a tempomandibular disorder pain screening (TMD) will be performed. Followed by the Nordic Orofacial Test Screening (NOT-S).

A Cone Beam CT (CBCT) scanning of the regions for implant placement will be performed using a Planmeca Viso 3D scanner; 100 kV, 12mA, voxel size 150 µm) with a FOV of 5 x 5 cm in both sides of the jaw for Kennedy class I dentition and in one side of the jaw for Kennedy class II dentitions.. This is estimated to give radiation of 2 x 50 µSv (Kennedy class 1 dentition) or 1 x 50 µSv, which is equivalent to a 7 hour t/r (Kennedy class 1 dentition) or a one way (Kennedy class 2 dentition) flight trip to New York in 10 km height.

T-scan (Tek-scan) and IOS-scan will be performed according to the description from the companies and OCA´s will be calculated.

Primary outcomes: Questionnaires on oral health and chewing Oral health Impact Profile 14, DC/TMD-screening test, Nordic Orofacial Screening test, Stellingsmas chewing ability questionnaire.

Secondary outcomes: Bite force and muscle strength Maximum bite force, tooth contact in intercuspal position, chewing time measurements and electromyography will be performed according to earlier descriptions.

The force during maximum tooth clenching will be recorded for 1 to 2 seconds with a strain-gauge transducer placed unilaterally on the mandibular first premolars. The transducer will be covered with protective plastic tubes and connected to an amplifier with peak storage facility. The molar bite force (N) will be assessed as the average of the stored peak values from right and left side (2 at each side with intervals of about 0.5 min).

EMG activity will be acquired bilaterally from the anterior temporal and masseter muscles during 1 to 2 seconds of maximal biting in the intercuspal position in 2 epochs with 1 min apart by means of a custom-designed 8-channel EMG system after amplification and filtering (gain 500-10,000; high-pass filter at 20-50 Hz and low pass at 1 kHz). The recordings will be performed with reusable, bipolar surface electrodes (tin plates, 3.0 x1.5 x 10.0 mm and 10-mm distance between electrodes) covered with electrode paste. After cleaning the skin with alcohol to reduce impedance, the electrodes will be placed transversely to the fiber direction.

Masticatory performance The chewing efficiency will be measured by the apple chewing time (seconds) as the duration of the chewing of a standardized slice of green, crisp apple (11 g Granny Smith with rind and core removed) from the first bite to the spontaneous termination swallow.

Also, the duration of the chewing cycle (milliseconds) during chewing of apple slices will be assessed by EMG from the average of 5 strokes in 2 chewing sequences measured automatically by the EMG system with the right anterior temporal muscle as reference muscle (definition of chewing cycle: from the start temporal activity of one closing phase to the start of temporal activity in the next closing phase).

Occlusal tooth contact The contact will be recorded clinically for all teeth and restorations. The contact was rated as 'firm' when the patient was able to maintain a straight plastic strip (0.05 x 6 mm) between the teeth against a strong pull, as 'near' contact if the strip could be pulled out but with resistance, and 'no' contact if there was no resistance to the pull. The contacts will be converted to occlusal units measures in premolar equivalent.

Ethical and data collection approval The project will be sent for approval at the local ethical committee. All procedures in the study will be conducted according to the 1964 Helsinki Declaration and its later amendments. Informed consent will be obtained from all participants included in the study on a written form approved by the Ethical Committee of the Medical Faculty at Copenhagen University. Participants will be informed about the risks of and alternatives to the proposed therapy.

Approval from Faculty of Health and Medical Sciences, Copenhagen University for processing of personal data (Case no 514-0798/23-3000).

Outcomes The primary clinical outcome of the first part of the study are OHRQoL measured with the validated Oral Health Impact Profile (OHIP-14) formula. It consists of 14 items rated in frequency on a Likert scale with five response options and according to score: very often (4), fairly often (3), occasionally (2), hardly ever (1), never (0) or don't know. Thus, an overall score between 0 and 56 can be obtained. A low score indicates good OHRQoL. The OHIP-14 patient questionnaire will be collected from the patients before and 1 month after the treatment with implant-supported crowns, bilaterally. Furthermore after 3- and 5-years follow-up.

The masticatory function in the first part of the study will be assessed with masticatory ability questionnaires and masticatory efficiency tests. Masticatory ability will be tested using the chewing ability questionnaire developed by Stellingsma and co-workers. In the questionnaire, the participants give their opinion about their ability to chew nine different kinds of food on a VAS scale. The items will be grouped into three scales A: soft food (boiled vegetables and potatoes, crustless bread, minced meat); B: tough food (crusty bread, steak, Gouda cheese) and C: hard food (apple, carrot, peanuts). The chewing time from putting the nine food items into the mouth and until swallowing will be measured in minutes and seconds with and without removable dental prosthesis (RDP) and 1 month after treatment with implant-supported crowns (ISC). The same intervals as above will be used for the bite force measurements and the occlusal contact area (OCA) (T-scan or Intraoral scanner) i.e., with (TRDP) and without (T0) RDPs and 1 month (T1) after treatment with ISC.

The maximum bite force will be measured using a U-shaped bite force transducer displaying force ranging from 0 -1000 (Kgf). The participants will be asked to clench their teeth for 5 s and the highest bite force displayed was noted as their peak value. The test will be repeated four times. Maximum bite force was measured initially in the session and the participants were given a two-minute rest before the next test was commenced.

In the second part of the study 2 digital methods for recording occlusal contacts will be examined and correlated to the conventional analog occlusal contacts registration with foils.

Occlusal contact area: The first method used to obtain an occlusal record will be the digital Tekscan (Tekscan Inc. Boston, MA). Each participant will be instructed in occlusion in the intercuspal occlusion position (IP) 3 times using maximum occlusal force and with a 100 my thick sensor foil placed in situ e.g., between the upper and lower jaw in IP. The T-scan software will generate a dynamic report showing an occlusal image of the relative bite force. One image of the 2D occlusal picture at maximum force and 2 other images at approximately 50% of the maximum force will be captured to compare occlusal registration at different clenching levels. The force will be determined by using a bite force measurement (Bite force equipment, Oslo, Norway) in the first premolar area. Each image will be coded and analyzed using computer software (Image J, NIH, US).

The second method of occlusal contact area will be assessed using a 3D intraoral digital scanner (IOS). Teeth in the maxillary and mandibular dental arch will be scanned intraorally and the relationship between the jaws will be registered by scanning the intercuspal occlusal position in both sites of the jaws. The IOS software will capture the scans and 2D pictures of the occlusal picture by normal intercuspal force (approximately half of the maximum bite force). An occlusal view of the 3D models will be selected, and the software will be programmed for automatic selection of the occlusal contact area (OCA).

The third method of describing the mandible jaw contact to the maxillary jaw is by occlusal units measured in premolar equivalent. This quite simple method is the most frequently used in the clinic. With 28 teeth the subject can have 18 occlusal pairs as the molars counts for two premolars. Clear shim stock foils are placed between the teeth and occlusal contact selection is based on an operator´s "resistance feel", when pulling the foil out from opposing occluding teeth. This is also called a static occlusal indicator and is the conventional method for occlusal contact registrations.

The third part of the study will compare splinted versus non-splinted crowns in a randomized design. Whether the crowns will be splinted or not are decided by distant randomization separate from clinicians conducting the trial. Twenty sealed envelopes will be opened where its stands whether the crowns has to be splinted crowns or non-splinted crowns. The implants in the splinted side will have an intermediate titanium abutment and impression will be taken at abutment level, whereas impressions in the non-splinted side will be taken directly at the fixture level. The splinted as well as the non-splinted crowns will be screw-retained and produced in monolithic zirconia. An open-tray technique / (scanning) will be used for both reconstructions.

The implant-supported reconstructions will be examined 1 month after insertion (baseline examination) and at 1-, 3- and 5-years follow-up examinations. At the baseline the former described methods for oral function and oral OHRQoL will be done, and biological and technical variables will be added. Marginal fit as well as other quality parameters of the reconstruction will be evaluated with the Copenhagen index score as well as an accessibility for oral hygiene score, Bleeding on probing (BOP), modified Gingival and plaque index as well and the incidence of mechanical complications including screw loosening's and ceramic chippings will be undertaken at baseline, 1-, 3- and 5-years follow-up examinations.

The marginal bone level will be evaluated at intraoral radiographs at the same intervals using customized radiographic positioning jigs to obtain periodically "identical" radiographs. Changes in marginal bone level (marginal bone loss, MBL) will be measured and calculated, and MBL will be the primary outcome variable for this part of the study.

Statistical analysis Using a significance level of 5% and a power of 90% with an improvement in Oral Health Related Quality of Life (OHIP-14) for 80% of the participants, (OHIP-14 change score > 2) the study will need 18 subjects. With a drop-out of five, 23 subjects in the upper or lower jaw are endeavored.

The data will be presented descriptively using mean and standard deviations to clarify small differences and to make comparison with other studies. Difference between groups in the outcome variables over time will be analyzed with linear mixed model. The tests will be performed by a statistician using the statistical program R and/or SPSS statistical software. A p-value of 0.05 or lower will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous subjects with missing posterior teeth (Kennedy class I or class II) in the upper or lower jaw, in need for fixed implant-supported crowns to replace the missing teeth are offered to be enrolled if they fulfill the following inclusion criteria. The participants must be in good health and with no contraindications for undergoing dento-alveolar surgery.

Exclusion Criteria:

* Untreated or active, progressive periodontitis
* Intake of (high dose) antiresorptive medicine or earlier medication related osteonecrosis of the jaw
* Therapeutic radiation to the head and neck
* Uncontrolled diabetes or systemic corticosteroids
* Heavy smoking (>20 cigarettes/day)
* An inability to open the mouth wide enough to place implants
* Decayed or unrestored anterior/premolar teeth
* Need for major bone augmentation (e.g., bone block graft, extensive augmentations with second operation for implant insertion)
* < 8 mm bone height to the alveolar nerve or sinus maxillaris
* Parafunctional habits or untreated temporomandibular dysfunctions or orofacial pain
* Unable to cooperate or too ill to complete the experiment
* Lack of signed informed consent

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Oral Health Related Quality of Life score | Up to 5 years
Oral Function change in percentage | Up to 5 years
Marginal Bone Loss in mm | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health and Medical Sciences, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided